CLINICAL TRIAL: NCT06156878
Title: Radiotherapy Combined With PD-1 Inhibitor and Anti-EGFR Monoclonal Antibody for Locally Advanced Nasopharyngeal Carcinoma Resistant to Induction Chemotherapy: A Prospective Phase II Study
Brief Title: PD-1 Inhibitor Plus Anti-EGFR Therapy And Radiotherapy in Locally Advanced NPC Resistant to Induction Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoshen Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022007
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; PD-1 inhibitor; Anti-EGFR monoclonal antibody; Induced chemotherapy resistance
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-EGFR and PD-1 inhibitor arm (Experimental): Two cycles of TP (docetaxel+cisplatin), TPF(docetaxel+cisplatin+5-FU), TPX (docetaxel+cisplatin+capecitabine) or GP regimen (gemcitabine+cisplatin) followed by radiotherapy (66-70.4Gy) combined with PD-1 inhibitor (every 3 weeks) and anti-EGFR monoclonal antibody (every 1 week) when responses to induction chemotherapy are less than 50% Partial Response (PR) or EBVDNA copy number decreased by less than 50%.
  Interventions: Combination Product: Anti-EGFR and PD-1 inhibitor arm

INTERVENTIONS:
Combination Product: Anti-EGFR and PD-1 inhibitor arm — Drug: PD-1 inhibitor and anti-EGFR monoclonal antibody The patients will receive radiotherapy (66-70.4Gy) combined with PD-1 inhibitor (every 3 weeks) and anti-EGFR monoclonal antibody (every 1 week). The specific treatment description is included in arm description.

SUMMARY:
Because nasopharyngeal carcinoma （NPC）is very sensitive to radiation and the specificity of the anatomical structure, radiotherapy has become the core treatment for NPC. Although induction chemotherapy combined with cisplatin-based concurrent chemoradiotherapy can effectively improve the overall survival and progression-free survival of NPC, such a sequential pattern can further exacerbate the toxic side effects of treatment, such as mucosal reactions and gastrointestinal toxicity. Therefore, it is particularly important to explore another treatment mode with high efficiency and low toxicity. Secondly, patients with poor response after induction chemotherapy indicate chemotherapy resistance. Whether patients can still benefit from concurrent platinum-based chemotherapy in the followed radiotherapy is doubtful. PD-1 inhibitor and anti-EGFR monoclonal antibody have proved to improve outcomes of head and neck cancers including EBV-related NPC, which have also showed relatively low toxicity. In this study, radiotherapy combined with PD-1 inhibitor and anti-EGFR monoclonal antibody were applied to treat patients with locally advanced NPC who were resistant to induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed locally advanced NPC; IHC EGFR positive; Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; Imaging assessment of MR after induction chemotherapy revealed the responses to induction chemotherapy are less than 50% Partial Response(PR) or EBVDNA copy number decreased by less than 50%; No prior anti-tumor treatment; Normal complete blood count; Normal hepatic function; Normal renal function (creatinine ≤ 1.5 times the upper limit of normal). -

Exclusion Criteria:

Previous radiotherapy; A history of any other type of malignancy; Pregnancy or lactation; Allergy to anti-EGFR monoclonal antibody; IHC EGFR negative; Allergy to PD-1 inhibitor; Obvious disfunction of liver, renal, cardiac or lung function; Un controlled infection; Systemic metastasis or distant metastasis; Patients with severe gastrointestinal diseases; Patients with mental disorders affecting patient participation in trial judgement; Cannot take contrast-MRI imaging.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  Progression Free Survival
OS | 3 years
  Overall Survival

SECONDARY OUTCOMES:
DCR | 3 years
  Disease-free survival
Number and percentage of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and RTOG | 3 years
  The detail number and percentage of adverse events by every systems Assessed by CTCAE v5.0 and RTOG.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China